CLINICAL TRIAL: NCT05653986
Title: A Prospective, Observational Diary Study to Evaluate the Real-World Effectiveness of the Acute Treatment of Migraine With Ubrogepant, When Used in Combination With Atogepant for Prevention
Brief Title: An Observational Study to Assess Change in Disease Activity When Ubrogepant Tablets Are Combined With Atogepant Tablets to Treat Migraine in Adult Participants
Acronym: COURAGE II
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-495
Record Dates: First submitted 2022-12-14; First posted 2022-12-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Migraine
Keywords: Migraine; Ubrogepant; Ubrelvy; Atogepant; Qulipta
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ubrogepant + Atogepant: Participants will receive ubrogepant in combination with atogepant as prescribed by their physician in routine clinical practice.

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will how effective the combination use of ubrogepant and atogepant is in treating adult participants with migraine. Change in migraine activity will be assessed.

Urogepant (Ubrelvy) and Atogepant (Qulipta) are approved drugs for treatment of migraine in adults in the US. Approximately 432 adult participants who are prescribed Ubrogepant and atogepant by their doctors will be enrolled in this study in the United States.

Participants will receive ubrogepant oral tablets and atogepant oral tablets as prescribed by their physician. Participants will be followed for 30 days.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Reports meeting migraine diagnostic criteria consistent with International Classification of Headache Disorders (ICHD) (i.e., they report symptoms accompanying their headaches that meet migraine criteria22 at screening).
* Currently using ubrogepant for acute treatment of migraine.
* Experienced at least 3 migraine attacks in the last 30 days.
* Currently taking atogepant for preventive treatment of migraine and has been taking atogepant, at the same dose, for at least 30 days.

Exclusion Criteria:

* Report currently taking Rimegepant (Nurtec®) for migraine treatment (acute or preventive).
* Report currently taking any of the anti-CGRP mAbs for preventive treatment of migraine:

  * Erenumab (Aimovig®)
  * Galcanezumab (Emgality®)
  * Fremanezumab (Ajovy®)
  * Eptinezumab (Vyepti®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with migraine using Migraine Buddy mobile application and prescribed Ubrogepant and Atogepant by their physician
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2022-12-18 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Meaningful Pain Relief | Up to approximately 30 days
  Meaningful relief occurs when the level of headache pain has been reduced to a degree that is meaningful to the participant; this can, but does not necessarily, occur prior to pain freedom. Participants will provide responses for ubrogepant-treated migraine attacks about the time to achieve meaningful relief of headache pain. This will result in a binary responder definition coded as "yes" for those achieving meaningful pain relief or "no" for those not satisfying that definition.
Percentage of Participants Who Return to Normal Function | Up to approximately 30 days
  Participants will also rate the ability to perform daily activities at the point when ubrogepant was taken using the Functional Disability Scale. The responses include "No disability (able to function normally)," "Mildly impaired (can still do everything but with difficulty)," "Moderately impaired (unable to do some things)," "Severely impaired (unable to do all or most things, bed rest may be necessary)." This will result in a binary responder definition coded as "yes" for those achieving return to normal function or "no" for those not satisfying that definition.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Montefiore/Albert Einstein /ID# 252243, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-495